CLINICAL TRIAL: NCT04278573
Title: Efficacy of Intralesional Vitamin D Injection for Treatment of Common Warts: A Randomized Controlled Trial
Brief Title: Intralesional Vitamin D Injection for Treatment of Common Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen P. Merry (Other)
Responsible Party: Sponsor-Investigator, Stephen P. Merry, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-010219
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 Treatment Group (Experimental): Subjects will receive a Vitamin D3 injection into their wart
  Interventions: Drug: Vitamin D3
- Placebo Group (Placebo Comparator): Subjects will receive a placebo injection into their wart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Intralesional injection of 0.3 ml 40,000 IU/ml vitamin D3 into one wart
  Other Names: Cholecalciferol
  Arms: Vitamin D3 Treatment Group
Drug: Placebo — 0.3 ml injection of sterilized sesame oil with no active study ingredient
  Arms: Placebo Group

SUMMARY:
Researchers are trying to find out if injecting Vitamin D into a wart is an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients seen at the Mayo Clinic Rochester practices
* Patients suffering from one or more cutaneous warts as diagnosed by the examining physician at baseline visit on typical diagnostic characteristics
* Able to provide consent
* Both recalcitrant and non-recalcitrant warts will be included

Exclusion Criteria:

* Patients with prior use of home or office-based destructive treatments for this wart(s) in the last 1 month with salicylic acid (SA) or cryotherapy
* Immunoadjuvant therapy for warts in the last 4 months (e.g Candida)
* History of vitamin D injection of warts ever
* High-dose vitamin D supplementation (>4,000 IU daily or equivalent) in the preceding 3 months
* Pregnancy or lactation
* Facial or genital warts
* Lesions not felt by the examining clinician to be a wart (e.g., corns or calluses)
* Immunosuppression (to include immunosuppressive medications or conditions as judged by the physician evaluating the patient at the baseline visit).
* Allergy to sesame oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Merry, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merry SP, Brennan DN, Duvall MJ, Stanek JB, O'Dowd EK, Thacher TD. Intralesional Injection of Vitamin D3 for Treatment of Cutaneous Warts: A Randomized, Double-Blind, Placebo-Controlled Trial. J Prim Care Community Health. 2025 Jan-Dec;16:21501319251365853. doi: 10.1177/21501319251365853. Epub 2025 Aug 23. PMID 40847834
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 Treatment Group | Placebo Group
Started | 41 | 36
Completed | 41 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 41 | 36 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (11.0) | 33.6 (10.1) | 35.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 41 | 34 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 36 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 36 | 77

OUTCOME MEASURES:

1. Primary Outcome: Complete Regression of Wart
Description: Number of subjects to have a complete resolution of cutaneous wart
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 36
Participants | 12 | 10

2. Secondary Outcome: Regression of Wart at 4 Weeks
Description: Number of participants who experienced complete regression of cutaneous wart at 4 weeks.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 36
Participants | 2 | 2

3. Secondary Outcome: Regression of Wart at 8 Weeks
Description: Number of participants who experienced complete regression of cutaneous wart at 8 weeks.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 36
Participants | 4 | 7

4. Secondary Outcome: Regression of Wart at 12 Weeks
Description: Number of participants who experienced complete regression of cutaneous wart at 12 weeks.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 Treatment Group | Placebo Group
Number analyzed (Participants) | 41 | 36
Participants | 7 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from the time of first injection of the investigational product until 112 days following the last administration of the investigational product, for a total of approximately 6 months.
Arm/Group | Vitamin D3 Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/36
Other Adverse Events (participants affected / at risk) | 41/41 | 36/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 Treatment Group (N=41) | Placebo Group (N=36)
Skin redness at injection site (General disorders) | 15 (15) | 15 (15)
Itching (General disorders) | 19 (19) | 19 (19)
Hematoma (blood blister) (General disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT04278573/Prot_SAP_000.pdf